CLINICAL TRIAL: NCT05177094
Title: Randomized, Placebo-Controlled, Phase 2 Clinical Trial to Evaluate LY3526318 for the Treatment of Diabetic Peripheral Neuropathic Pain
Brief Title: Chronic Pain Master Protocol (CPMP): A Study of LY3526318 in Participants With Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17597; H0P-MC-NP02 (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-01-03; First posted 2022-01-04 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3526318 (Experimental): Participants received 250 milligram (mg) of LY3526318 orally, once daily for the first 4 weeks and were switched to placebo once daily for the next 4 weeks of the treatment period.
  Interventions: Drug: LY3526318
- Placebo (Placebo Comparator): Participants received placebo orally, once daily, for 8-weeks treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3526318 — Administered orally
  Arms: LY3526318
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and efficacy of study drug LY3526318 for the treatment of diabetic peripheral neuropathic pain (DPNP). This trial is part of the chronic pain master protocol H0P-MC-CPMP (NCT05986292) which is a protocol to accelerate the development of new treatments for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Have a visual analog scale (VAS) pain value ≥40 and <95 during screening.
* Have a history of daily pain for at least 12 weeks based on participant report or medical history.
* Have a body mass index <40 kilograms per meter squared (kg/m²) (inclusive).
* Are willing to maintain a consistent regimen of any ongoing nonpharmacologic pain-relieving therapies (for example, physical therapy) and will not start any new nonpharmacologic pain-relieving therapies during study participation.
* Are willing to discontinue all pain medications taken for chronic pain conditions for the duration of the study.
* Have daily symmetrical foot pain secondary to peripheral neuropathy present for at least 6 months and as diagnosed through use of the Michigan Neuropathy Screening Instrument Part B ≥3 (©University of Michigan).
* Have a history and current diagnosis of type 1 or type 2 diabetes mellitus.
* Have stable glycemic control as indicated by a glycated hemoglobin ≤11 at time of screening.
* Are men, or women able to abide by reproductive and contraceptive requirements.

Exclusion Criteria:

* Have had a procedure within the past 6 months intended to product permanent sensory loss in the target area of interest (for example, ablation techniques).
* Have surgery planned during the study for any reason, related or not the disease state under evaluation.
* Have, in the judgment of the investigator, an acute, serious, or unstable medical condition or a history or presence of any other medical illness that would preclude study participation.
* Have a substance use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (5th edition; DSM-5; American Psychiatric Association).
* Have had cancer within 2 years of baseline, except for cutaneous basal cell or squamous cell carcinoma resolved by excision.
* Have fibromyalgia
* Are, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.
* Have a positive human immunodeficiency virus (HIV) test result at screening.
* Have an intolerance to acetaminophen or paracetamol or any of its excipients.
* Have a history of alcohol, illicit drug, analgesic or narcotic use disorder within 2 years prior to screening.
* Have a current drug-induced neuropathy, for example, due to some types of chemotherapy, or other types of peripheral neuropathy.
* Have known hereditary motor, sensory or autonomic neuropathies.
* Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (35):
  - Synexus Clinical Research US, Inc., Chandler, Arizona
  - Synexus Clinical Research - Glendale, Glendale, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Alliance for Multispecialty Research, LLC Tempe, Tempe, Arizona
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - CMR of Greater New Haven, Hamden, Connecticut
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Suncoast Research Group, Miami, Florida
  - University of Miami Don Suffer Clinical Research Building, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus Clinical Research US, Inc - Orlando, Orlando, Florida
  - Synexus Clinical Research US, Inc., Pinellas Park, Florida
  - Synexus Clinical Research US, Inc - Orlando, The Villages, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Synexus Clinical Research US, Inc., Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Skokie, Illinois
  - Boston Clinical Trials, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Synexus - Cincinnati, Cincinnati, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - FutureSearch Trials, Austin, Texas
  - Cedar Health Research, Dallas, Texas
  - Synexus - US, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Puerto Rico (2):
  - Ponce Medical School Foundation Inc., Ponce
  - Latin Clinical Trial Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Chronic Pain Master Protocol (CPMP): A Study of LY3526318 in Participants With Diabetic Peripheral Neuropathic Pain — https://trials.lillytrialguide.com/en-US/trial/1L5jVzms1JQf2Av5xg5rrU

RESULTS

PARTICIPANT FLOW:
Groups:
- 250 Milligram (mg) LY3526318: Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks and were switched to placebo once daily for the next 4 weeks of the treatment period.
Period: Overall Study
Arm/Group | 250 Milligram (mg) LY3526318 | Placebo
Started | 103 | 52
Received at Least One Dose of Study Drug (Safety Population Week 1-4) | 102 | 52
Safety Population Week 5-8 (All participants who took at least 1 dose of study drug and who did not discontinue at or prior to week 4.) | 95 | 46
Completed | 88 | 43
Not Completed | 15 | 9
Not completed — Adverse Event | 5 | 5
Not completed — Non-compliance With Study Drug and Procedures | 0 | 1
Not completed — Protocol Deviation | 3 | 0
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Participant could not tolerate long study visits | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 250 mg LY3526318: Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks and were switched to placebo once daily for the next 4 weeks of the treatment period.
- Total: Total of all reporting groups
Arm/Group | 250 mg LY3526318 | Placebo | Total
Number analyzed (Participants) | 103 | 52 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 26 | 80
  >=65 years | 49 | 26 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.3) | 63.6 (8.1) | 63.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 27 | 69
  Male | 61 | 25 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 6 | 14
  White | 90 | 42 | 132
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 2 | 0 | 2
  United States | 101 | 52 | 153
Average Pain Intensity as Measured by the Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: score on a scale] — The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  score on a scale | 5.80 (1.87) | 5.99 (1.68) | 5.87 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Pain Intensity as Measured by the Numeric Rating Scale (NRS)
Description: The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine. Posterior mean change from baseline, 95 percent (%) credible intervals was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: All enrolled participants who took at least 1 dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 94 | 46
score on a scale | -1.50 [-1.81 to -1.19] | -1.35 [-1.80 to -0.90]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.15, 95% CI 2-sided [-0.70 to 0.40] — Posterior mean difference with 95% credible interval is reported

2. Primary Outcome: Change From Baseline in Average Pain Intensity as Measured by the Numeric Rating Scale (NRS)
Description: The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine. Posterior mean change from baseline, 95% credible intervals was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: All enrolled participants who took at least 1 dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 85 | 38
score on a scale | -1.80 [-2.17 to -1.42] | -1.78 [-2.32 to -1.24]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.01, 95% CI 2-sided [-0.66 to 0.64] — Posterior mean difference with 95% credible interval is reported

3. Secondary Outcome: Change From Baseline in the Brief Pain Inventory-Short Form Modified (BPI-SFM) Total Pain Interference Score
Description: The BPI-SFM is a numeric rating scale that assesses the severity of pain (severity scale) and its impact on daily functioning (Pain Interference scale). BPI-SFM pain interference scale has been reported here. Pain interference scale has 7 items, including general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life each assessed on a 10-point scale. All the 7-items are averaged to produce a total score ranging from 0 to 10 where, 0=does not interfere to 10=completely interferes and the mean is reported here. Higher score represents worse outcome. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 47
score on a scale | -1.54 [-1.90 to -1.17] | -1.41 [-1.90 to -0.91]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.13, 95% CI 2-sided [-0.72 to 0.46] — Posterior mean difference with 95% credible interval is reported

4. Secondary Outcome: Change From Baseline in the Brief Pain Inventory-Short Form Modified (BPI-SFM) Total Pain Interference Score
Description: as for outcome 3
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 44
score on a scale | -1.69 [-2.14 to -1.25] | -1.43 [-2.05 to -0.81]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.26, 95% CI 2-sided [-0.98 to 0.46] — Posterior mean difference with 95% credible interval is reported

5. Secondary Outcome: Change From Baseline for Overall Improvement as Measured by Patient's Global Impression of Change
Description: Patients Global Impression of change captured the participant's perspective of treatment apart from sub-aspects of the general improvement. This is a numeric scale from 1 to 7: 1=very much better, and 7=very much worse. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 47
score on a scale | 2.77 [2.55 to 3.00] | 2.99 [2.67 to 3.31]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.22, 95% CI 2-sided [-0.61 to 0.18] — Posterior mean difference with 95% credible interval is reported

6. Secondary Outcome: Change From Baseline for Overall Improvement as Measured by Patient's Global Impression of Change
Description: as for outcome 5
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 44
score on a scale | 2.77 [2.54 to 3.01] | 2.94 [2.61 to 3.28]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.17, 95% CI 2-sided [-0.58 to 0.24] — Posterior mean difference with 95% credible interval is reported

7. Secondary Outcome: Change From Baseline for Worst Pain Intensity as Measured by NRS
Description: The NRS was used to describe pain severity. Participants were asked to describe their worst pain over the past 24 hours, on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 94 | 46
score on a scale | -1.48 [-1.81 to -1.15] | -1.36 [-1.83 to -0.88]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.12, 95% CI 2-sided [-0.68 to 0.45] — Posterior mean difference with 95% credible interval is reported

8. Secondary Outcome: Change From Baseline for Worst Pain Intensity as Measured by NRS
Description: as for outcome 7
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 85 | 38
score on a scale | -1.68 [-2.09 to -1.26] | -1.74 [-2.32 to -1.14]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.06, 95% CI 2-sided [-0.65 to 0.77] — Posterior mean difference with 95% credible interval is reported

9. Secondary Outcome: Change From Baseline on the Visual Analog Scale (VAS) for Pain
Description: VAS was a graphic, single-item scale where participants were asked to describe their pain intensity over the past week, on a scale of 0 to 100: 0=no pain, and 100=worst imaginable pain. Participants completed the VAS by placing a line perpendicular to the VAS line at a point that described their pain intensity. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 47
score on a scale | -21.84 [-26.33 to -17.38] | -18.75 [-24.99 to -12.55]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -3.09, 95% CI 2-sided [-10.43 to 4.28] — Posterior mean difference with 95% credible interval is reported

10. Secondary Outcome: Change From Baseline on the Visual Analog Scale (VAS) for Pain
Description: as for outcome 9
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 44
score on a scale | -23.11 [-28.31 to -17.95] | -21.61 [-28.74 to -14.50]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -1.50, 95% CI 2-sided [-10.04 to 7.00] — Posterior mean difference with 95% credible interval is reported

11. Secondary Outcome: Change From Baseline on the Sleep Scale From the Medical Outcomes Study (MOS Sleep Scale) - Average Hours of Sleep
Description: The MOS Sleep Scale consists of 12 questions addressing the past week. Question 1 asks time to fall asleep and it is reported in 5-point timeframe categories. Question 2 asks average hours of sleep. In the remaining 10 questions participants report how often a sleep symptom or problem was present on a scale ranging from '0=all of the time' to '5=none of the time.' MOS Sleep scale dimension scores range from 0 to 100 with lower score indicating improvement, except for the dimension of sleep adequacy, where higher scores indicate improvement. Here, the average hours of sleep (i.e., Question 2) is reported as the average number of hours slept each night during the past week (range 0 to 24 hours). Higher number of hours slept indicates improvement. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: hours per night
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 47
hours per night | 0.40 [0.14 to 0.66] | 0.29 [-0.07 to 0.65]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.12, 95% CI 2-sided [-0.32 to 0.54] — Posterior mean difference with 95% credible interval is reported

12. Secondary Outcome: Change From Baseline on the Sleep Scale From the Medical Outcomes Study (MOS Sleep Scale) - Average Hours of Sleep
Description: as for outcome 11
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: hours per night
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 44
hours per night | 0.45 [0.17 to 0.74] | 0.25 [-0.13 to 0.63]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.20, 95% CI 2-sided [-0.24 to 0.65] — Posterior mean difference with 95% credible interval is reported

13. Secondary Outcome: Total Amount of Rescue Medication Use as Measured by Average Daily Dosage
Description: Total amount of rescue medication use as measured by average daily dosage. Posterior mean, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg per day (mg/day)
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 94 | 46
mg per day (mg/day) | 255.71 [163.50 to 347.62] | 211.35 [81.10 to 342.14]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 44.36, 95% CI 2-sided [-114.73 to 204.00] — Posterior mean difference with 95% credible interval is reported

14. Secondary Outcome: Total Amount of Rescue Medication Use as Measured by Average Daily Dosage
Description: as for outcome 13
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/day
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 85 | 38
mg/day | 138.75 [62.87 to 215.62] | 237.51 [126.82 to 346.84]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -98.76, 95% CI 2-sided [-231.86 to 34.49] — Posterior mean difference with 95% credible interval is reported

15. Secondary Outcome: Change From Baseline on the EuroQuality of Life Five Dimensions (5D) Five Level (5L) Questionnaire (EQ-5D-5L) Health State Index (United States Algorithm)
Description: The EQ-5D-5L assessed quality of life based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant was asked to 'check the ONE box that best describes your health TODAY,' choosing from 5 options (no problems, slight problems, moderate problems, severe problems, extreme problems) provided under each dimension. The scores in the 5 dimensions were summarized into a health state index score using the United States algorithm. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than dead) with higher scores indicating better health: 0=a health state equivalent to death, and 1=perfect health.
  Posterior mean change from baseline, 95% credible intervals was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 47
score on a scale | 0.04 [-0.00 to 0.08] | 0.03 [-0.02 to 0.09]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.01, 95% CI 2-sided [-0.05 to 0.07] — Posterior mean difference with 95% credible interval is reported

16. Secondary Outcome: Change From Baseline on the EuroQuality of Life Five Dimensions (5D) Five Level (5L) Questionnaire (EQ-5D-5L) Health State Index (United States Algorithm)
Description: as for outcome 15
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 44
score on a scale | 0.05 [-0.01 to 0.10] | 0.05 [-0.02 to 0.13]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.01, 95% CI 2-sided [-0.09 to 0.08] — Posterior mean difference with 95% credible interval is reported

ADVERSE EVENTS:
Time Frame: Baseline through Week 8
Description: All participants under the safety population for week 1-4 and week 5-8.
Groups:
- 250 mg LY3526318 Week 1-4: Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks of treatment period (Week 1-4).
- 250 mg LY3526318/Placebo Week 5-8: Participants who received 250 mg of LY3526318 in the first 4 weeks were switched to received placebo once daily for the next 4 weeks of the treatment period (Week 5-8).
- Placebo Week 1-4: Participants received placebo orally, once daily, for week 1 to 4 of treatment period.
- Placebo Week 5-8: Participant from Week 1-4 continued to receive placebo orally, once daily, for week 5 to 8 of treatment period.
Arm/Group | 250 mg LY3526318 Week 1-4 | 250 mg LY3526318/Placebo Week 5-8 | Placebo Week 1-4 | Placebo Week 5-8
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/95 | 0/52 | 0/46
Serious Adverse Events (participants affected / at risk) | 2/102 | 3/95 | 1/52 | 1/46
Other Adverse Events (participants affected / at risk) | 40/102 | 23/95 | 22/52 | 10/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg LY3526318 Week 1-4 (N=102) | 250 mg LY3526318/Placebo Week 5-8 (N=95) | Placebo Week 1-4 (N=52) | Placebo Week 5-8 (N=46)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg LY3526318 Week 1-4 (N=102) | 250 mg LY3526318/Placebo Week 5-8 (N=95) | Placebo Week 1-4 (N=52) | Placebo Week 5-8 (N=46)
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 2 | 1
Fatigue (General disorders) | 3 | 0 | 2 | 1
Covid-19 (Infections and infestations) | 1 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 5 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 4 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0
Medical device site irritation (General disorders) | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 2 | 0 | 0
Lymphocyte count (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Poor quality sleep (Psychiatric disorders) | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 3 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT05177094/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT05177094/SAP_001.pdf